CLINICAL TRIAL: NCT01354587
Title: Evaluation of Efficacy and Tolerability of Hizentra® in Subjects Transitioning From Vivaglobin® (16% SCIG Product) to Hizentra® (20% SCIG Product)
Brief Title: Evaluation of Efficacy and Tolerability of Hizentra®
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hizentra
Record Dates: First submitted 2011-03-18; First posted 2011-05-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Primary Immunodeficiency Disorders
Keywords: immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Immunologic Deficiency Syndromes | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hizentra (Active Comparator): Compare IgG levels and site reaction in subjects transitioning from Vivaglobin to Hizentra
  Interventions: Drug: Hizentra

INTERVENTIONS:
Drug: Hizentra — Subjects transition from Vivaglobin to Hizentra using weekly subcutaneous infusions for 32 weeks.

SUMMARY:
The purpose of this study is to measure the changes in the Treatment Satisfaction Questionnaire for Medication in the areas of effectiveness, side effects, and convenience of administration of each medication in Primary Immunodeficiency Disorder (PIDD) subjects transitioning from subcutaneous Vivaglobin® to Hizentra®.

DETAILED DESCRIPTION:
This trial will evaluate subjects with Primary Immunodeficiency Disorder (PIDD) who are currently self-infusing Vivaglobin therapy for at least six months prior to changing to Hizentra® therapy. Following screening and enrollment, subjects will continue to self-infuse Vivaglobin® for seven infusions and then be converted to subcutaneous Hizentra® treatment which they will continue for the next 6 months. The study will determine if Hizentra® provides improved subject satisfaction by Treatment Satisfaction Questionnaire for Medication. Diaries related to the local site reactions, the number of infusion sites per subject/per dose, volume of Hizentra® per site, duration of infusions, systemic side effects of the new medication and dose on IgG levels and antibody titers, and local site reactions with Hizentra®.

ELIGIBILITY:
Inclusion Criteria:

* Subjects currently self-infusing with Vivaglobin® for at least six months prior to enrollment.
* Diagnosis of antibody deficiency due to primary immune deficiency disease.
* Stable serum IgG levels of > 550 mg/dl while on Vivaglobin® based on two determinations at least 8 weeks apart and obtained within 6 months of entry.
* Willing to sign consent and follow study schedule.
* 1 year to 75 years of age.

Exclusion Criteria:

* Evidence of acute systemic illness or infection at within four weeks of screening or enrollment.
* Any serious grade 3 or greater toxicity at screening.
* History of bleeding or chronic skin disorders.
* Selective IgA deficiency in absence of other antibody deficiencies
* History of anaphylactic or severe systemic reaction to Vivaglobin.
* Pregnant or breastfeeding females.
* Use of systemic pre-medication prior to SCIG.
* Protein losing enteropathy or nephritic syndrome.
* Any condition that in the opinion of the investigator would interfere with the conduct of the study.
* Subject or guardian unwilling to sign consent or adhere to study schedule.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To measure the changes in the Treatment Satisfaction Questionnaire for Medication in PIDD subjects transitioning from subcutaneous Vivaglobin® to Hizentra®. | 32 weeks
  Subjects complete the TSQM at each study visit

SECONDARY OUTCOMES:
To compare the incidence of local site reactions in subjects self-infusing with Vivaglobin® transitioning to Hizentra®. | 32 weeks
  Study subjects complete a weekly infusion diary that is collected at each study visit.
To compare the steady state IgG levels in subjects self-infusing with Vivaglobin® transitioning to Hizentra®. | 32 weeks
  IgG levels are obtained at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: John Sleasman, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, St. Petersburg, Florida, United States